CLINICAL TRIAL: NCT05569369
Title: Endovascular Management of Combined Common Femoral and Superficial Femoral Arteries Lesions in Patients With Chronic Lower Limb Threatening Ischemia
Brief Title: Endovascular Management of Combined Common Femoral and Superficial Femoral Arteries Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Eldin AHmed Soliman, Hossam Eldin Ahmed Soliman Mohamed, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-23
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Lower Limb Ischemia
MeSH Terms: interventions — Angioplasty; Stents; Atherectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- angioplasty with stenting (Experimental)
  Interventions: Procedure: angioplasty and stenting

INTERVENTIONS:
Procedure: angioplasty and stenting — dilatation of stenotic arteries and insertion of stent
  Other Names: atherectomy

SUMMARY:
The purpose of this study is to evaluate the technical feasibility, safety, and 1-year clinical efficacy of the endovascular treatment of patients with atherosclerotic common femoral artery (CFA) obstructions with associated superficial femoral artery lesions. Participants will undergo angioplasty with or without stenting of common femoral and superficial femoral arteries.

DETAILED DESCRIPTION:
Study design:

It is a prospective study which will include patients who need revascularization after approval of this study from local ethical committee and obtaining written informed consent.

Study setting:

This study will be done in Sohag University Hospitals and in Cairo University Hospitals.

Study sample:

This study will include 25 patients who present with chronic lower limb threatening ischemia and need endovascular revascularization and met the eligible criteria.

All patients in the study are subjected to the following: - (A) History

Complete history taking from all patients with special concern of the following:

* Age, sex and life style.
* History of diabetes, hypertension, dyslipidemia, stroke and coronary artery disease.
* History of smoking, congestive heart failure and chronic renal disease.
* History of blood diseases and hypercoagulable states.
* History of local or systemic infection.
* History of previous revascularization in the same limb and the other limbs. (B)Examination

General examination:

* General condition.
* Vital signs: - (pulse, blood pressure, temperature, respiration).
* Systemic examination and preoperative medical assessment especially cardiopulmonary and renal systems evaluation.

Local examination:

* Examination of the arterial pulsation all over the arterial tree.
* Measuring ankle brachial index (ABI) and toe brachial index (TBI).
* Examination of any wound and measuring its dimensions. (c) Investigation Including: _
* Complete blood count, lipid profile, fasting blood sugar and HgA1C.
* Bleeding time and coagulation time.
* Prothrombin time and concentration, serum urea and creatinine.
* Echocardiography and ECG.
* Arterial duplex of the affected limb.
* CT angiography of abdominal aorta and both lower limbs unless creatinine clearance (CrCl) is impaired (D) Procedure All procedures will be performed in the operating room by vascular surgeons. Local anesthesia with conscious sedation is indicated, unless general anesthesia is needed in patients who are restless and in pain.

Access to the lesion is achieved either by way of an over-the-aortic bifurcation approach with the use of a dedicated 6-F or 7-F-long sheath (45 cm) or via a brachial approach with the use of a dedicated 6-F or 7-F-long sheath (90 cm) or retrograde via popliteal approach if failed antegrade approach.

After sheath placement, an intravenous bolus of 50 UI kg-1 of heparin is given. Digital subtraction angiography (DSA) is performed to assess lesions. After successful passage of the target lesions with a hydrophilic 0.035-inch guide wire, primary stenting without lesion pre-dilatation is preferably performed. One stenting technique from the CFA to the superficial femoral artery (SFA) may be involved.

The last generation of self-expandable stents eg The Supera stent will be used in common femoral artery lesions.

Balloon-expandable stents are used for associated SFA lesions. Self-expandable stents are routinely post-dilated. The balloon dimensions are chosen such that the nominal diameter is inferior to the stent diameter by 1 mm to reduce medial damage and the length doesn't exceed the stent length. The technical result of the procedure is assessed by DSA.

A prophylactic dose of low-molecular-weight heparin is given during the duration of hospitalization to prevent venous thrombo-embolic events. Postoperatively, patients are prescribed aspirin (75-160 mg day-1) and clopidogrel (75 mg day-1) for 6 months. After 6 months, patients are prescribed only clopidogrel (75 mg day-1).

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine < 2.
* Complaining of chronic lower limb threatening ischemia due to denovo atherosclerotic disease i.e. no previous intervention of common femoral artery with associated superficial femoral artery lesion (Rutherford stages 2-5).

Exclusion Criteria:

* - Non-atherosclerotic conditions (for example: vasculitis, collagen vascular disease, Buerger's disease, radiation).
* Acute limb ischemia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
sustained clinical improvement. | 1 year
  a sustained upward shift of ≥1 category of the Rutherford classification without the need for repeated target lesion revascularization in surviving patients.

IPD SHARING:
Plan to Share IPD: No